CLINICAL TRIAL: NCT07186465
Title: Evaluating Urinary Microbiome Modulation :An RCT of Antibiotic vs Gynoflor Prophylaxis in Postmenopausal Women With Recurrent Cystitis
Brief Title: Microbiome-Modulating Prophylaxis RCT: Antibiotic vs Gynoflor in Postmenopausal Women With Recurrent Cystitis
Acronym: microbiome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MURA2024/339; Ref.2024/671 (Other: HREC, Ramathibodi Hospital, Mahidol Univ.)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cystitis, Recurrent; Urinary Tract Infections
Keywords: Postmenopausal Women; Nitrofurantoin; Antibiotic Prophylaxis; Gynoflor; Lactobacillus; Estriol; Vaginal Probiotics; Urinary Microbiome; 16S rRNA Sequencing; qPCR; Lower Urinary Tract Symptoms; RUTISS Questionnaire; Adherence Monitoring; Antimicrobial Resistance; Thailand
MeSH Terms: conditions — Cystitis; Recurrence; Urinary Tract Infections; Lower Urinary Tract Symptoms | interventions — Nitrofurantoin

STUDY DESIGN:
Intervention Model Description: Randomized, two-arm, parallel-group, open-label trial in postmenopausal women with recurrent UTI. Participants are allocated 1:1 by computer-generated block randomization to: (a) nitrofurantoin 100 mg orally at bedtime for 6 months, or (b) Gynoflor vaginal tablet nightly for 14 days then twice weekly through month 6. Baseline and month-6 clinic visits with labs/microbiome sampling; twice-weekly remote check-ins for adherence, symptoms, and AEs. If symptomatic UTI occurs, treat per standard care and then continue assigned prophylaxis to complete 6 months.
Masking Description: Open-label study; no masking of participants, care providers, investigators, or outcomes assessors. Allocation is revealed at randomization. Blinding is not feasible because the interventions differ in route and schedule (oral nitrofurantoin vs vaginal Lactobacillus/estriol). Laboratory analyses (urine culture, qPCR, 16S rRNA) use coded sample IDs to reduce bias, but allocation could be accessed if needed; therefore the study is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrofurantoin Prophylaxis (Active Comparator): Nightly oral nitrofurantoin 100 mg for 6 months as prophylaxis for recurrent UTI in postmenopausal women. If symptomatic UTI occurs, treat per standard care and, once resolved, continue assigned prophylaxis to complete 6 months. Monitoring per protocol: baseline and month-6 visits with urinalysis, urine culture, urinary microbiome, and kidney function; twice-weekly phone/Line check-ins for adherence, symptoms, and adverse events.
  Interventions: Drug: Nitrofurantoin
- Gynoflor Vaginal Tablet (Experimental): Vaginal tablet containing Lactobacillus with ultra-low-dose estriol (Gynoflor) for 6 months: insert 1 tablet nightly for 14 days, then twice weekly through month 6. Same monitoring and management as comparator: if UTI occurs, treat per standard care and then resume assigned prophylaxis to finish 6 months.
  Interventions: Drug: Gynoflor

INTERVENTIONS:
Drug: Nitrofurantoin — Nightly oral nitrofurantoin 100 mg for 6 months as prophylaxis for recurrent UTI in postmenopausal women. If symptomatic UTI occurs, treat per standard care and, once resolved, continue assigned prophylaxis to complete 6 months. Monitoring per protocol: baseline and month-6 visits with urinalysis, urine culture, urinary microbiome, and kidney function; twice-weekly phone/Line check-ins for adherence, symptoms, and adverse events.
  Other Names: Nitrofurantoin macrocrystals/monohydrate
  Arms: Nitrofurantoin Prophylaxis
Drug: Gynoflor — Vaginal tablet containing Lactobacillus with ultra-low-dose estriol. Insert 1 tablet nightly for 14 days, then twice weekly through month 6 as prophylaxis against recurrent urinary tract infection. If a symptomatic UTI occurs, treat per standard of care; after resolution, continue assigned prophylaxis to complete 6 months. Monitoring identical to comparator.
  Other Names: Vaginal Lactobacillus with ultra-low-dose estriol
  Arms: Gynoflor Vaginal Tablet

SUMMARY:
This open-label, parallel-group randomized controlled trial compares two prophylaxis strategies for recurrent urinary tract infection (rUTI) in postmenopausal women: (1) nightly oral nitrofurantoin 100 mg for 6 months versus (2) a vaginal tablet containing Lactobacillus with ultra-low-dose estriol (Gynoflor: nightly for 14 days, then twice weekly to month 6). Participants (≥40 years) are randomized 1:1 in computer-generated blocks and followed for 6 months. The primary endpoint is the proportion with rUTI recurrence within 6 months. Secondary endpoints include time to first recurrence, antibiotic resistance in breakthrough infections, change in lower urinary tract symptoms (Thai RUTISS), and urinary microbiome measures (Lactobacillus dominance and community diversity by qPCR and 16S rRNA). Key assessments occur at baseline and month 6 (urinalysis, culture, urinary microbiome sampling, and kidney function). Adherence and adverse events are captured via twice-weekly phone/Line contacts. Approximately 100 participants (50 per arm) will be enrolled as a feasibility-sized pilot.

DETAILED DESCRIPTION:
Background and Rationale

Recurrent cystitis is common after menopause and burdens quality of life and healthcare use. Antibiotic prophylaxis is effective but may promote antimicrobial resistance with long-term use. Vaginal Lactobacillus with ultra-low-dose estriol can restore urogenital flora and potentially reduce rUTI and lower urinary tract symptoms. Comparative data versus nightly antibiotic prophylaxis-and effects on the urinary microbiome-remain limited. This trial directly evaluates clinical recurrence and microbiome modulation with nitrofurantoin versus a Lactobacillus/estriol vaginal tablet over 6 months.

Objectives

Primary objective: Compare the 6-month rUTI recurrence proportion between nitrofurantoin and Gynoflor.

Key secondary objectives: (a) time to first recurrence; (b) antimicrobial resistance patterns in breakthrough infections; (c) change in Thai RUTISS score; (d) Lactobacillus dominance and within-sample diversity of the urinary microbiome.

Key Endpoint Definitions

rUTI recurrence (primary): ≥1 symptomatic episode meeting clinical criteria with urine culture growth of a uropathogen during the 6-month follow-up (episodes during temporary treatment holds still count toward the endpoint).

Time to first recurrence: days from randomization to first qualifying rUTI.

Antibiotic resistance: susceptibility profile of cultured uropathogens from breakthrough infections, categorized per local laboratory standards.

Microbiome metrics: quantitative Lactobacillus abundance (qPCR) and alpha diversity indices from 16S rRNA profiling.

Design Overview

Open-label, two-arm, parallel RCT with 1:1 allocation by concealed, computer-generated block randomization. Follow-up is 6 months. Masking is not feasible due to intervention routes; laboratory personnel for microbiome and culture testing are shielded from allocation where practicable.

Interventions (Summary)

Nitrofurantoin arm: 100 mg orally once nightly through month 6.

Gynoflor arm: one vaginal tablet nightly for 14 days, then twice weekly (e.g., Monday/Friday) through month 6.

(Rescue treatment for symptomatic UTI follows standard of care; study prophylaxis resumes afterward to complete 6 months.)

Study Procedures (Selected)

Baseline (Day 0): consent, randomization, Thai RUTISS, urinalysis, urine culture, urinary microbiome sampling, BUN/creatinine.

Follow-up (Months 0-6): twice-weekly phone/Line check-ins to reinforce adherence and capture symptoms/adverse events; prompt clinical evaluation if UTI symptoms arise.

Month 6: repeat Thai RUTISS, urinalysis/culture, urinary microbiome sampling, BUN/creatinine.

Specimen handling: midstream clean-catch urine; UA ~20 mL, culture 5-10 mL, microbiome ~50 mL. Samples processed promptly or refrigerated at 4 °C ≤24 h if needed.

Laboratory Methods (Overview)

Urinary microbiome assays are performed at the Department of Medical Sciences: (1) qPCR estimating Lactobacillus abundance across time points; (2) 16S rRNA gene sequencing for community profiling and alpha diversity.

Sample Size and Analysis Plan (Pilot)

Approximately 100 participants (50/arm) are planned based on local feasibility for an initial pilot. Analyses will follow intention-to-treat with supportive per-protocol summaries. The primary endpoint will be compared between arms using a risk difference with 95% CIs and a chi-square or Fisher's exact test. Time-to-event data will be presented with Kaplan-Meier estimates and log-rank testing. Continuous outcomes (e.g., Thai RUTISS change) will use t-tests or Wilcoxon rank-sum as appropriate; paired pre/post within-arm changes will use paired tests. Missing outcome data will be handled by complete-case analysis with sensitivity analyses (e.g., worst-case imputation for the primary endpoint) if missingness >5-10%.

Safety Monitoring and Adherence

Expected risks include nitrofurantoin intolerance (e.g., GI upset, hypersensitivity), local vaginal irritation, minor phlebotomy discomfort, and time burden. Adverse events are solicited during twice-weekly contacts and at visits; serious adverse events are reported per IRB policy. Given the low-risk profile and pilot scope, a formal DSMB is not planned; the PI and study team review safety at regular intervals. Adherence is promoted by structured reminders and documented via participant report during check-ins.

Data Management and Quality

Case report forms are source-verified against electronic medical records and laboratory outputs. Microbiome and culture laboratories follow internal QC procedures; analytical staff are kept unaware of allocation when feasible. Randomization files are access-restricted; analysis is pre-specified prior to database lock.

ELIGIBILITY:
Inclusion Criteria:

* Female, postmenopausal, age ≥40 years
* Clinical history of recurrent urinary tract infection (rUTI) as assessed by the investigator
* Able and willing to take assigned prophylaxis for 6 months
* Able to attend baseline and Month 6 study visits and provide urine samples
* Able to provide written informed consent
* Willing and able to complete twice-weekly phone/LINE follow-ups

Exclusion Criteria:

* Current symptomatic UTI at enrollment (may be treated and reconsidered after resolution)
* Known hypersensitivity or contraindication to nitrofurantoin or to the Lactobacillus/estriol vaginal tablet (Gynoflor) or their excipients; significant renal impairment or other label-based contraindications to nitrofurantoin per local practice
* Planned urologic surgery or procedure expected during the 6-month study period
* Recent bacterial vaginosis (e.g., within the past month) or active vulvovaginal skin disorders precluding vaginal product use
* History of hormone-dependent malignancy (e.g., breast, uterine, or cervical cancer) or unexplained abnormal vaginal bleeding
* Significant liver disease (e.g., active hepatitis) or other conditions judged by the investigator to make participation unsafe
* Participation in another interventional trial that could interfere with outcomes
* Withdrawal of consent or severe adverse event requiring discontinuation

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with recurrent UTI within 6 months | Baseline to 6 months after randomization
  Number of participants who experience ≥1 episode of symptomatic urinary tract infection (UTI) during the 6-month prophylaxis period, confirmed by clinical symptoms and positive urine culture per hospital standard. Event counted once per participant; groups compared between arms.

SECONDARY OUTCOMES:
Time to first recurrent UTI | Baseline to 6 months
  Days from randomization to first symptomatic, culture-confirmed UTI during the 6-month period; participants without an event are censored at 6 months.
Antibiotic resistance among breakthrough infections | During the 6-month prophylaxis period
  Proportion of bacterial isolates from breakthrough UTIs that are non-susceptible to commonly tested antibiotics per local microbiology reporting.
Change in lower urinary tract symptom score (RUTISS, Thai) | Baseline and month 6
  Change in Recurrent Urinary Tract Infection Symptom Scale (RUTISS) Section C Severity Score
  Description: Mean change in the Recurrent Urinary Tract Infection Symptom Scale (RUTISS) Section C total severity score from baseline to Month 6. Section C summarizes four domains (urinary symptoms, urinary presentation, UTI pain/discomfort, bodily sensations). The Overall RUTISS Severity Score is calculated as: sum of Section C responses ÷ 11 × 10, yielding a 0-100 scale. Higher scores = worse symptom/pain severity.
  Time Frame: Baseline and Month 6.
  Unit of Measure: Points (0-100).
  Scale Details: Minimum = 0, Maximum = 100, Higher = worse
Lactobacillus abundance by qPCR | Baseline and month 6
  Change in Lactobacillus copy number/relative abundance in midstream urine measured by quantitative PCR.
Urinary microbiome diversity by 16S rRNA sequencing | Baseline and month 6
  Change in alpha-diversity indices of urine microbiota profiles determined by 16S rRNA gene sequencing.
Incidence of adverse events related to intervention | Up to 6 months
  Number and proportion of participants with any intervention-related adverse event
Adherence to assigned prophylaxis | During 6 months
  Proportion of scheduled doses taken, assessed by medication logs and twice-weekly contacts

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital Mahidol University, Bangkok, Phayatai Ratchathewi, Thailand

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome results will be shared. A data dictionary and coding key will be provided. Direct identifiers will be removed and dates shifted as needed. Data will be shared for research purposes only and not for commercial use.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available beginning 12 months after the primary results are published (or 24 months after database lock, whichever comes first) and for 5 years thereafter.
Access Criteria: Qualified researchers may request access by emailing the study PI/central contact with: (1) a brief proposal and analysis plan, (2) documentation of ethics/IRB approval or exemption, and (3) a signed Data Use Agreement. Requests will be reviewed by the study steering team. Approved users will receive data via secure transfer; re-identification attempts and onward sharing are prohibited, and publications must acknowledge the original study.